CLINICAL TRIAL: NCT07233785
Title: Comparison of the Postoperative Analgesic Efficacy of the Combination of Adductor Canal Block and Biceps Femoris Short Head Block Versus Adductor Canal Block Alone in Patients Undergoing Total Knee Arthroplasty
Brief Title: Comparison of ACB With ACB and BiFeS Combination in Knee Arthroplasty Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2025-09/52
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain Management; Knee Surgery; Knee Arthroplasty, Total
Keywords: postoperative pain; knee arthroplasty; biceps femoris short head; bifes; adductor canal blok; regional anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor Canal Block (Active Comparator): For an adductor canal block, a high-frequency ultrasound probe will be placed on the anterior aspect of the patient's thigh, approximately at the midpoint between the inguinal crease and the medial condyle of the knee. (The depth is generally 3-5 cm). Using an in-plane technique, the needle will be advanced from lateral to medial, passing through the sartorius or vastus medialis muscle, and 20 mL of 0.25% bupivacaine will be injected around the femoral artery.
  Interventions: Procedure: Adductor Canal Block (ACB) Only
- Combination of Adductor Canal Block and Biceps Femoris Short Head Block (Active Comparator): For adductor canal block, a high-frequency ultrasound probe will be placed on the anterior aspect of the patient's thigh, approximately at the midpoint between the inguinal crease and the medial condyle of the knee. (The depth is generally 3-5 cm). Using in-plane technique, the needle passing through the sartorius or vastus medialis muscle, and 20 mL of 0.25% bupivacaine will be injected around the femoral artery.
  For BiFeS block, a high-frequency ultrasound probe will be placed on the distal posterior aspect of the thigh. The Biceps Femoris Short Head (BiFeS) muscle will be visualized at the distal lateral part of the femur, near the lateral supracondylar line, and the needle tip will be placed at the interface between the BiFeS and the lateral supracondylar line of the femur. 20 mL of 0.25% bupivacaine will be injected, and during the injection, it will be confirmed by ultrasound that the solution lifts the muscle and spreads along the bone surface.
  Interventions: Procedure: Adductor Canal Block (ACB) + Biceps Femoris Short Head Block (BiFeS)

INTERVENTIONS:
Procedure: Adductor Canal Block (ACB) Only — 20 mL of 0.25% bupivacaine
  Arms: Adductor Canal Block
Procedure: Adductor Canal Block (ACB) + Biceps Femoris Short Head Block (BiFeS) — 20 mL of 0.25% bupivacaine
  Arms: Combination of Adductor Canal Block and Biceps Femoris Short Head Block

SUMMARY:
The aim is to compare the postoperative analgesic effects of Adductor Canal and Biceps Femoris Short Head Blocks with Adductor Canal Block in patients undergoing Knee Arthroplasty surgery

DETAILED DESCRIPTION:
Patients were divided into two randomized groups: Group 1 (ACB group, n=30) and Group 2 (ACB+BiFeS group, n=30). All patients will receive the same standard spinal anesthesia per hospital protocol. All blocks will be applied with the same ultrasonography and block equipment, and by the same physician. After the surgery, patients in Group 1 will receive Adductor Canal Block (ACB) with 20 mL of 0.25% bupivacaine. Patients in Group 2 will receive Adductor Canal Block with 20 mL of 0.25% bupivacaine and Biceps Femoris Short Head (BiFeS) with 20 mL of 0.25% bupivacaine. Routine analgesic procedure consisting of 3x400mg Ibuprofen will be followed postoperatively for 24 hours. Numeric Rating Scale (NRS) will be used to assess postoperative pain on 1st, 6th, 12th, 18th and 24th hours after the surgery. Tramadol 1mg/kg IV will be administered as a rescue analgesic for all patients if NRS score is higher than 4. Total Tramadol consumption will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age who underwent percutaneous nephrolithotomy under general anesthesia and were I-II-III according to the American Society of Anesthesiologists (ASA) risk classification were included in the study.

Exclusion Criteria:

* patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with known allergies to any of the study drugs,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment
* patients who wanted to withdraw from the study,
* patients with alcohol and drug addiction,
* patients with musculoskeletal abnormalitie

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-10-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
1. Numeric Rating Scale (NRS) Scores | Postoperative 24 hours
  Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Total tramadol consumption | Postoperative 24 hours
  Postoperative total analgesic need was recorded as "milligram" in unit.

CONTACTS AND LOCATIONS:
Overall Officials: OĞUZ GÜNDOĞDU, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation; BUĞRA KARATAŞ, Study Chair — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No